CLINICAL TRIAL: NCT01180712
Title: Study of Oral Anthocyanins on Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC 10/S0802/27; Rowett 901 (Other: Rowett institute study code)
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes
Keywords: anthocyanin; blaeberries; bilberries; blueberries; mirtoselect; type 2 diabetes; insulin resistance; Adipose tissue; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blaeberry concentrated caspule (Active Comparator): 30 obese male subjects (BMI > 30) with type 2 diabetes controlling their diabetes by diet alone or impaired glucose tolerance.
  Volunteers will be given a total daily dose of 1.4 grams of mirtoselect (a concentrated blaeberry extract) a day formulated in hard gelatin capsules (0.47 gram per capsule) administered thrice a day for 21 days.
  Mirtoselect provided by Indena S.p.A. (http://www.mirtoselect.info/)
  Interventions: Dietary Supplement: Mirtoselect
- Placebo capsules containing lactose (Placebo Comparator): 30 obese male subjects (BMI > 30) with type 2 diabetes controlling their diabetes by diet alone or impaired glucose tolerance.
  Volunteers will be given a placebo consisting of lactose formulated in hard gelatin capsules administered thrice a day for 21 days.
  Interventions: Dietary Supplement: Mirtoselect

INTERVENTIONS:
Dietary Supplement: Mirtoselect — Male subjects (BMI > 30) with type 2 diabetes controlling their diabetes by diet alone or impaired glucose tolerance.
  Volunteers will be given either a total daily dose of 1.4 grams of concentrated blaeberry extract (mirtoselect provided by Indena S.p.A. (http://www.mirtoselect.info/) in a hard gelatin capsules or control capsules containing lactose administered thrice a day for 21 days.

SUMMARY:
Dietary strategies for alleviating the metabolic complications such as diabetes associated with obesity are actively being pursued as alternatives to pharmaceutical interventions The genus Vaccinium (e.g. blueberry, blaeberry, cranberry) has been used traditionally as a source of folk remedies for established diabetic symptoms, primarily as leaf or stem infusions or decoctions. Berries from this family such as blaeberry (BL) and blueberry (BB) are enriched in anthocyanins, polyphenolics recognized for their ability to provide and activate cellular antioxidant protection, inhibit inflammatory gene expression, and consequently protect against oxidant-induced and inflammatory cell damage and cytotoxicity. The association of obesity with adipose tissue stress, macrophage recruitment, and inflammatory gene expression suggests that eating edible berries from this genus might provide an effective alternative or supplementary intervention to attenuate obesity- associated inflammation and the associated insulin resistance.

The aim of this study is to determine the effects of anthocyanin supplementation in the form of a concentrated blaeberry extract on insulin resistance and inflammation particularly in the adipose tissue following a three week supplementation period.

ELIGIBILITY:
Inclusion Criteria:

* Obese male subjects (BMI > 30)
* Aged > 40 and < 70 years of age
* Type 2 diabetes; subjects controlling their diabetes by diet alone or with impaired glucose tolerance
* All the obese subjects will have a waist circumference over 40 inches
* All subjects must live the Aberdeenshire area of Scotland

Exclusion Criteria:

Medical exclusion criteria:

* Chronic illness, including:

  * thromboembolic or coagulation disease,
  * unregulated thyroid disease,
  * kidney disease,
  * hepatic disease,
  * severe gastrointestinal disorders,
  * pulmonary disease (e.g. chronic bronchitis, COPD),
* Alcohol or any other substance abuse,
* Eating disorders,
* Psychiatric disorders (including severe depression, lithium treatment, schizophrenia, severe behavioural disorders),
* Skin conditions on the abdomen,
* Allergy to skin dressings,

Medication exclusion criteria:

* Oral steroids,
* Tricyclic antidepressants, neuroleptics,
* Anticoagulants,
* Digoxin and antiarrhythmics,
* Chronic use of antiinflammatories (e.g. high doses of aspirin, ibuprofen),
* Insulin, Sulphonylureas, Thiazolidinediones (glitazones), metformin

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Oral Glucose Tolerance Test | Day 0 and 21 days post intervention
  Change in Oral Glucose Tolerance following intervention

SECONDARY OUTCOMES:
Fasting blood glucose/insulin | Day 0, 7, 14, and 21 days post intervention
  Change in fasting blood glucose/insulin in response to intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hoggard, PhD, Principal Investigator — University of Aberdeen Rowett Institute of Nutrition and Health
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, United Kingdom

REFERENCES:
- [Background] Martineau LC, Couture A, Spoor D, Benhaddou-Andaloussi A, Harris C, Meddah B, Leduc C, Burt A, Vuong T, Mai Le P, Prentki M, Bennett SA, Arnason JT, Haddad PS. Anti-diabetic properties of the Canadian lowbush blueberry Vaccinium angustifolium Ait. Phytomedicine. 2006 Nov;13(9-10):612-23. doi: 10.1016/j.phymed.2006.08.005. Epub 2006 Sep 18. PMID 16979328
- [Background] Zafra-Stone S, Yasmin T, Bagchi M, Chatterjee A, Vinson JA, Bagchi D. Berry anthocyanins as novel antioxidants in human health and disease prevention. Mol Nutr Food Res. 2007 Jun;51(6):675-83. doi: 10.1002/mnfr.200700002. PMID 17533652
- [Background] Lau FC, Bielinski DF, Joseph JA. Inhibitory effects of blueberry extract on the production of inflammatory mediators in lipopolysaccharide-activated BV2 microglia. J Neurosci Res. 2007 Apr;85(5):1010-7. doi: 10.1002/jnr.21205. PMID 17265471
- [Background] DeFuria J, Bennett G, Strissel KJ, Perfield JW 2nd, Milbury PE, Greenberg AS, Obin MS. Dietary blueberry attenuates whole-body insulin resistance in high fat-fed mice by reducing adipocyte death and its inflammatory sequelae. J Nutr. 2009 Aug;139(8):1510-6. doi: 10.3945/jn.109.105155. Epub 2009 Jun 10. PMID 19515743

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT01180712/Prot_SAP_000.pdf